CLINICAL TRIAL: NCT05281614
Title: Immune Effects of Vedolizumab With or Without Anti-TNF Pre-treatment in T1D
Acronym: COBRA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB22-007
Record Dates: First submitted 2022-02-17; First posted 2022-03-16 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2023-02

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Etanercept; vedolizumab

STUDY DESIGN:
Intervention Model Description: open label study with 2 treatment arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Arm A will receive 6 weeks of vedolizumab after 8 weeks of etanercept. Final study visit at 52 weeks.
  Interventions: Drug: Etanercept; Drug: Vedolizumab
- Arm B (Experimental): Arm B will receive 6 weeks of vedolizumab only. Final study visit at 52 weeks.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Etanercept — Etanercept is a fully humanized monoclonal antibody that targets TNFα.
  Other Names: Enbrel
  Arms: Arm A
Drug: Vedolizumab — Vedolizumab is a humanized monoclonal antibody that targets α4ß7 integrin.
  Other Names: Entyvio

SUMMARY:
The underlying hypothesis is that vedolizumab will modify immune cell trafficking in type 1 diabetes, and that this will be enhanced by pre-treatment with etanercept. This study will determine whether there is mechanistic evidence in support of this hypothesis and provide preliminary information about safety, efficacy, and tolerability of vedolizumab with and without pretreatment with etanercept in adults with type 1 diabetes (T1D)

DETAILED DESCRIPTION:
Vedolizumab directly blocks integrin α4ß7 on circulating immune cells preventing their egress from the blood, while etanercept blocks the TNFα signaling necessary for the α4ß7 cognate addressin MAdCAM-1 to be expressed in pancreatic endothelial cells. For these reasons, the investigators hypothesize that the two agents may synergistically prevent diabetogenic immune cells from trafficking from the periphery to their target tissue to cause islet cell destruction. Cells from both the myeloid (e.g., myeloid DC1 cells and non-classical monocytes) and lymphoid compartments (e.g., diabetes antigen-specific T cells) would be impacted by this therapeutic combination.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18-45 years of age, inclusive
2. Diagnosis of T1D between 21 days and 3 years from screening
3. Positive for at least one diabetes-related autoantibody any time since diagnosis, including but not limited to:

   * Glutamate decarboxylase (GAD-65)
   * mIAA, if obtained within 10 days of the onset of exogenous insulin therapy
   * IA-2
   * ZnT8 (Zinc transporter 8)
4. Random (non-fasting) C-peptide or peak MMTT stimulated C-peptide ≥ 0.2 pmol/mL.
5. Females of child-bearing potential must be willing to use effective birth control from the screening visit through 12 weeks post last dose of study medication.
6. Up to date for clinically recommended immunizations including COVID-19 and seasonal influenza vaccine at least 3 weeks prior to baseline treatment.
7. Willing to forgo live vaccines 6 weeks prior to baseline treatment visit until 6 weeks following last treatment visit.
8. HbA1c ≤ 8.5% at screening
9. Willing and able to give informed consent for participation

Exclusion Criteria:

1. History of severe reaction or anaphylaxis to human, humanized or murine monoclonal antibodies
2. History of malignancy or serious uncontrolled cardiovascular, nervous system, pulmonary, renal, or gastrointestinal disease
3. History of immunodeficiency
4. Recent (within 3 months) serious bacterial, viral, fungal, or other infections
5. Pending or positive SARS-CoV-2 test or symptoms of possible COVID-19 illness at baseline treatment visit.
6. Serologic evidence of current or past HIV, Hepatitis B, or Hepatitis C.
7. Positive QuantiFERON or PPD TB test, history of tuberculosis, or active TB infection.
8. Active infection with EBV as defined by real-time polymerase chain reaction (PCR).
9. Active infection with CMV as defined by real-time PCR.
10. Clinically significant liver function abnormalities as defined by ALT or AST> 1.5 x the upper limit of age-determined normal (ULN).
11. Any of the following hematologic abnormalities:

    * White blood count <3,000/μL or >14,000/μL
    * Lymphocyte count <800/μL
    * Platelet count <75,000 /μL
    * Hemoglobin <10.0 g/dL
    * Neutrophil count <1500 cells/μL
12. Females who are pregnant or lactating.
13. Receipt of live vaccine (e.g., varicella, MMR (measles, mumps and rubella), intranasal influenza vaccine) within 6 weeks of randomization.
14. Receipt of other vaccines within 3 weeks of baseline treatment.
15. Receipt of an immune modulating biologic or investigational drug within 3 months or 5 half-lives before screening visit.
16. Use of non-insulin therapies aimed to control hyperglycemia within 30 days of screening visit.
17. History of other clinically significant autoimmune disease needing chronic therapy with biologics or steroids with the exception of celiac disease and stable thyroid disease.
18. Use of medications known to influence glucose tolerance. Topical, nasal, inhaled corticosteroids acceptable per investigator discretion.
19. Any medical or psychological condition that in the opinion of the principal investigator would interfere with the safe completion of the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Impact on insulin secretion determined by 2-hour MMTT stimulated AUC C-peptide 10 weeks after first vedolizumab dose and 52 weeks after randomization. | baseline dose to 10 weeks and baseline dose to 52 weeks
  MMTT-Stimulated 2-Hour C-peptide AUC is the mean area under the C-peptide level time curve over the 2-hour period divided by the duration after a mixed-meal tolerance test.
Adverse events of etanercept treatment as a measure of safety and tolerability | baseline to 52 weeks
  An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. Results will be reported as a rate of each adverse event
Adverse events of vedolizumab treatment as a measure of safety and tolerability | baseline to 52 weeks
  An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. Results will be reported as a rate of each adverse event

SECONDARY OUTCOMES:
Frequency of α4β7+ T cells | baseline to 52 weeks
  Cell phenotype will be measured as a percentage using either flow cytometry or cytometry by time of flight (CyTOF), via an assay such as the AIM (Activation-Induced Marker) assay.
Frequency of myeloid DC1 cells | baseline to 52 weeks
  Cell phenotype will be measured as a percentage using either flow cytometry or cytometry by time of flight (CyTOF), via an assay such as the AIM (Activation-Induced Marker) assay.
Frequency and surface marker phenotype of other immune cells such as antigen specific CD4 and CD8 cells, memory and naive T and B cells | baseline to 52 weeks
  Cell phenotype will be measured as a percentage using either flow cytometry or cytometry by time of flight (CyTOF), via an assay such as the AIM (Activation-Induced Marker) assay.
Change in T1D antibody titers | baseline to 52 weeks
  T1D autoantibodies include: mIAA, GAD-65, IA-2, ZnT8, as reported in international units per mililiter

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California San Diego, La Jolla, California
  - Benaroya Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided